CLINICAL TRIAL: NCT03277677
Title: The Effect of Fluid Resuscitation With 0.9% Sodium Chloride Versus Balanced Crystalloid Solution on Renal Function of Sepsis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Nattachai Srisawat ,M.D., Associated professor, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB.113/60
Record Dates: First submitted 2017-09-07; First posted 2017-09-11 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Sepsis; Septic Shock; Acute Kidney Injury
MeSH Terms: conditions — Sepsis; Shock, Septic; Acute Kidney Injury | interventions — Saline Solution; Ringer's acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- normal saline (Active Comparator)
  Interventions: Drug: Normal saline
- balanced solution (Active Comparator)
  Interventions: Drug: Ringer's Acetate

INTERVENTIONS:
Drug: Normal saline — for resuscitation in sepsis patients
  Arms: normal saline
Drug: Ringer's Acetate — for resuscitation in sepsis patients
  Arms: balanced solution

SUMMARY:
The high chloride content of 0.9%sodium chloride (0.9%NaCl) leads to adverse pathophysiological effects in both animals and healthy human volunteers. Small randomized trials confirm that the hyperchloremic acidosis induced by 0.9%NaCl also occurs in patients. A strong signal is emerging from recent large propensity-matched and cohort studies for the adverse effects that 0.9% NaCl has on the clinical outcome in surgical and critically ill patients when compared with balanced crystalloids. Major complications are the increased incidences of acute kidney injury and the need for renal replacement therapy, and that pathological hyperchloremia may increase postoperative mortality.

Fluid resuscitation with 0.9% NaCl in animals with sepsis resulted in hyperchloremic metabolic acidosis, worsened AKI, and increased mortality when compared with resuscitation with a balanced crystalloid solution.

Furthermore, hyperchloremic acidosis also resulted in increased concentrations of circulating inflammatory mediators in an experimental model of severe sepsis in rats, with a dose-dependent increase in circulating interleukin-6, tumor necrosis factor-a, and interleukin-10 concentrations with increasing acidosis.

Thus, in this study, investigators compared the effects of a balanced crystalloid solution with 0.9% NaCl on the renal function in severe sepsis/septic shock patients. Investigators hypothesized that balanced crystalloid solution resuscitation would decrease AKI incidence and severity and would improve immunomodulatory effect when compared with 0.9% NaCl resuscitation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Who need fluid resuscitation in the Emergency Room (ER).
* Who have fulfilled the criteria for sepsis/septic shock within the previous 24 hours according to sepsis is defined as life-threatening organ dysfunction caused by a dysregulated host response to infection.

  o Patients with infection and resulted from a host's systemic inflammatory response syndrome (SIRS) to infection are defined as sepsis if meet the criteria 2 or more of
  * Temperature >38°C or <36°C
  * Heart rate >90/min
  * Respiratory rate >20/min or PaCo2 <32 mm Hg (4.3 kPa)
  * White blood cell count >12000/mm3 or <4000/mm3 or >10% immature bands.
* Patient who have Septic shock is a subset of sepsis in which underlying circulatory and cellular/metabolic abnormalities are profound enough to substantially increase mortality.

  o Patients with septic shock can be identified with a clinical construct of sepsis with persisting hypotension requiring vasopressors to maintain MAP ≥65 mm Hg and having a serum lactate level >2 mmol/L (18 mg/dL) despite adequate volume resuscitation.
* AND where informed consent is obtainable either from the patient or by proxy (first degree relative, spouse) if patients aren't in fully conscious status (eg.comatose, drowsiness, irritable).

Exclusion criteria

Exclusion Criteria:

* Patients with chronic kidney disease (CKD) defined by baseline serum creatinine > 2.0 in male and 1.5 in female.
* Patients with End stage renal disease (ESRD) with or without renal replacement therapy.
* Patients with active cardiac disease : severe valvular heart, cardiomyopathy, decompensated heart failure NYHA II-IV, severe pulmonary hypertension.
* HIV/AIDs Patients.
* Allergy towards 0.9% NaCl or Ringer's Acetate.
* Any form of renal replacement therapy.
* Intracranial bleeding within current hospitalization.
* Therapy with corticosteroid or non steroidal anti-inflammatory substance.
* Patients who predicted not to survive more than 24 hours.
* Pregnant and lactating patients.
* Withdrawal of active therapy.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
The incidence of acute kidney injury for any stage and severity | at day 7

SECONDARY OUTCOMES:
The neutrophil function (chemotaxis, CD11b ) between two randomized groups at | 0, 24, and 72 hours after resuscitation.
The monocyte function (HLA-DR) between two randomized groupsafter resuscitation. | at 0, 24, and 72 hours after resuscitation.
The inflammatory marker (IL-6, IL-10) between two randomized groups at | 0, 24, and 72 hours after resuscitation.
Urinary neutrophil gelatinase-associated lipocalin (NGAL) after randomization and after resuscitation with trial fluid | at 0,24 and 72 hours after resuscitation.
Urinary liver-type fatty acid binding protein (L-FABP) | at 0,24 and 72 hours after resuscitation.
Sequential [Sepsis-related] Organ Failure Assessment (SOFA) Score. (excluding Glasgow Coma Score) at 72 hours after randomization. | at 72 hours after randomization.
Need of renal replacement therapy within 72 hours after randomization | within 72 hours after randomization
Days alive without renal replacement therapy | in 28 days after randomization
Hospital length of stay for survivors sanctioned | at 28 days after randomization

CONTACTS AND LOCATIONS:
Locations (1):
- Chulalongkorn university, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No